CLINICAL TRIAL: NCT05187052
Title: Rigid Telescopes, C-MAC, Flexible Bronchoscopy for Intubation in Patients With Anticipated Difficult Airways
Acronym: Rigidscopes
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Yaser Said Cetin, MD, Yuzuncu Yil University
Other Study IDs: VBEAK 2020/12-02
Record Dates: First submitted 2021-11-15; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Videolaryngoscopy
Keywords: Airway management, Difficult airway, Tracheal intubation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 (REI group): Group 1 included patients that were intubated using rigid endoscope-assisted orotracheal intubation (REI) (0°, 45°, and 70°), 18-cm rigid telescope (Storz, Germany), full-HD camera (Olympus, USA), and Macintosh blade.
  Interventions: Other: Tracheal intubation
- Group 2 (V-MAC Group): Group 2 included patients that underwent endotracheal intubation using a V-MAC (Besdata, China) videolaryngoscope and Magill forceps.
  Interventions: Other: Tracheal intubation
- Group 3 (FFEI group): Group 3 included patients that underwent flexible fiberoptic endotracheal intubation (FFEI Group, Storz, Germany).
  Interventions: Other: Tracheal intubation

INTERVENTIONS:
Other: Tracheal intubation — Video-assisted intubation technique

SUMMARY:
The primary outcome of the study is the first-attempt orotracheal intubation success rate and the secondary outcomes include intubation time, mucosal injury, and complications during intubation.

DETAILED DESCRIPTION:
Difficult airway management in phonomicrosurgery requiring endotracheal tube (ETT) placement is highly important for both the anesthetist and the surgeon. The use of rigid telescopes in the intubation of children with difficult intubation, such as those with Pierre Robin sequence (PRS), has been previously described in the literature. In addition, the use of Airtraq™ and rigid endoscopes in patients undergoing phonomicrosurgery, particularly in patients with difficult laryngoscopy, has also been reported in the literature. However, the uses of these techniques have mostly been described in the administration of surgery or in defining airway disease. In this study, we aimed to evaluate the use of rigid telescopes during intubation, particularly in patients with a difficult airway, and to compare them with videolaryngoscope Macintosh (V-MAC) and flexible fiberoptic bronchoscope.

ELIGIBILITY:
Inclusion Criteria:

Patients with a modified Cormack-Lehane (C-L) grade of 3 and 4, Wilson score of ≥ 6, Thyromental distance (TMD) distance of ≤ 6 cm, Sternomental distance (SMD) ≤ 13.

Exclusion Criteria:

Patients that had severe mouth opening (<2.5 cm), Required nasotracheal intubation, Upper airway and pharyngeal diseases, Presence of cervical spine anomalies, Emergency procedures, Failed mask ventilation, ASA III and IV score, Patients who were allergic to any of the drugs to be used during premedication and anesthesia.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Difficult airway management in phonomicrosurgery requiring endotracheal tube (ETT) between 18-90 years old patients.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of three video laryngoscopes: Rigid telescopes, C-MAC, flexible bronchoscopy for intubation in patients with anticipated difficult airways | 1 day
  Successful intubation at first attempt
Comparison of three video laryngoscopes: Rigid telescopes, C-MAC, flexible | 1 day
  Intubation time (sec)

SECONDARY OUTCOMES:
Comparison of three video laryngoscopes: Rigid telescopes, C-MAC, flexible | 1 day
  Labial mucosa injury, Dental injury, Oral and pharyngeal mucosal injury, Vocal cord or lesion injury,

CONTACTS AND LOCATIONS:
Locations (1):
- Yaser Said Cetin, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol